CLINICAL TRIAL: NCT05003245
Title: A Phase 3 Randomized Double-masked Active Controlled Study to Compare the Efficacy and Safety of HLX04-O Administered by Intravitreal Injection with Ranibizumab in Subjects with Wet Age Related Macular Degeneration (wAMD)
Brief Title: Compare the Efficacy and Safety of HLX04-O with Ranibizumab in Subjects with WAMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLX04-O-wAMD-CN
Record Dates: First submitted 2021-07-08; First posted 2021-08-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Vascular Endothelial Growth Factor A; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX04-O (Experimental): Biologic recombinant anti-VEGF humanized monoclonal antibody
  Interventions: Drug: HLX04-O，recombinant anti-vascular endothelial growth factor (VEGF) humanized monoclonal antibody ophthalmic injection
- Ranibizumab (Active Comparator): Biologic anti-VEGF recombinant humanized monoclonal antibody fragment
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: HLX04-O，recombinant anti-vascular endothelial growth factor (VEGF) humanized monoclonal antibody ophthalmic injection — 0.05mL solution at a 4-week interval for intravitreal injection
  Arms: HLX04-O
Drug: Lucentis — 0.05mL solution at a 4-week interval for intravitreal injection
  Arms: Ranibizumab

SUMMARY:
this study will compare the efficacy and safety of HLX04-O administered by IVT with ranibizumab in patients with active CNV secondary to AMD.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized double masked active controlled study to compare the efficacy and safety of HLX04-O administered by IVT with ranibizumab in patients with active CNV secondary to AMD. The study will be conducted in approximately 60 sites in China.

Either HLX04-O (1.25 mg) IVT or ranibizumab (0.5 mg) IVT will be administered at a 4-week interval for 1 year (12 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Capable to understand and sign the informed consent form (ICF) which includes compliance with the ICF and this protocol. In the Investigator's judgment, willing and able to complete all visits and assessments adhering to the prohibitions and restrictions specified in this protocol.
2. Women or men aged ≥50 years when signing the ICF.
3. Newly diagnosed, untreated, active subfoveal or juxtafoveal CNV lesions secondary to AMD in the study eye. (Active CNV was defined as leakage on FA and subretinal or intraretinal fluid on OCT with confirmation of the reading center during screening).
4. The total lesion area (including hemorrhage, scar and neovascularization) of the study eye ≤12 disc area (DA) with confirmation of the reading center before randomization a.
5. The BCVA letters between 24 and 73, inclusive, in the study eye, using Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
6. Clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm the diagnosis.
7. Participants' fellow (non-study) eye must have had a BCVA of 24 letters or better.

Exclusion Criteria:

1. Macular-related retinal pigment epithelial tears in the study eye; scar, fibrosis or atrophy involving the fovea, or CNV due to other causes in the study eye (e.g., ocular histoplasmosis, trauma, or pathological myopia etc.) with confirmation of the reading center.
2. The fellow (nonstudy) eye needs anti-VEGF IVT injection (e.g. CNV due to wAMD, trauma, pathological myopia, retina vein occlusion, diabetic macular edema, etc) in the next 3 months after randomization, in the investigator's judgment.
3. Active or recent (within 1 month prior to dose 1) intraocular, extraocular or periocular infection (including conjunctivitis, keratitis, scleritis or endophthalmitis), or history of idiopathic or autoimmune-associated uveitis in either eye.
4. Vitreous hemorrhage in the study eye within 3 months prior to dose 1.
5. Aphakia (except intraocular lens) or posterior capsular rupture of the lens (except yttrium aluminium-garnet (YAG) laser posterior capsulotomy after intraocular lens implantation ≥1 month prior to first dose) in the study eye.
6. Corneal dystrophy or history of corneal transplantation, scleral softening or history of scleral softening, history of rhegmatogenous retinal detachment or macular hole (Stage II, III or IV) in the study eye.
7. Uncontrolled glaucoma (defined as intraocular pressure [IOP] ≥25 mmHg despite treatment with antiglaucoma medication), and/or glaucoma filtering surgery (e.g., trabeculectomy, scleral nipping, non-penetrating trabeculectomy, etc.), or advanced glaucoma resulting in a cup/disc ratio >0.8 in the study eye
8. Equivalent spherical diopter of the study eye ≥-8D. For participants who had undergone refractive correction or cataract surgery, the equivalent spherical diopter of the study eye before surgery ≥-8D.
9. Estimated by the Investigator, any concurrent intraocular condition except wAMD (e.g., diabetic retinopathy, dry AMD, retina vein occlusion, uveitis, angioid streaks, retinal detachment, epiretinal membrane, amblyopia, central serous chorioretinopathy, etc.) in the study eye that limited the potential to gain visual acuity upon treatment with the investigational product, or could have required medical or surgical intervention during the study to prevent or treat visual loss.
10. Underwent intraocular surgery including verteporfin photodynamic therapy (PDT), transpupillary thermotherapy, macular translocation, vitrectomy, laser photocoagulation in macular area, other surgery in macular area or surgery to treat AMD.
11. Previous extraocular or periocular surgery within 1 month or intraocular surgery (including cataract surgery, etc.) within 3 months prior to dose 1, or current unhealed wound, moderate or severe ulcer or history of fracture in the study eye.
12. Subconjunctival or intraocular or systemic use of corticosteroids within 3 months (including subconjunctival or intraocular long-acting implant within 6 months) prior to dose 1 in the study eye.
13. Previous systemic anti-VEGF therapy or IVT injection of any anti-VEGF drug into either eye or other ocular use of anti-VEGF drug within 3 months prior to dose 1.
14. Participated in any drug (other than vitamins and minerals) or device clinical trials within 3 months or the duration of 5 half-lives of the study drug (which is longer) prior to dose 1 and have used the test drug or received device treatment.
15. Pregnancy or lactation.
16. Infertile women fail to meet either of the following ones: 1) menopause (≥12 continuous months of amenorrhea with no identified cause other than menopause before screening); 2) surgically sterilized.

    Men or fertile women fail to meet both of the following ones: 1) women of childbearing potential must have a negative urine or serum pregnancy test result within 14 days prior to initiation of the study intervention, and should not breastfeed; If the urine pregnancy test is positive, it must be confirmed by a serum pregnancy test; 2) agreement to remain abstinent (refrain from heterosexual intercourse) or use effective contraceptive methods from signed ICF to at least 6 months following the last dose of the study intervention. Effective contraceptive methods include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices (IUDs), and copper IUDs.
17. In the Investigator's judgment, there is evidence of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the participant at high risk for treatment complications (e.g. stroke or myocardial infarction within 6 months prior todose1, uncontrolled hypertension (systolic blood pressure≥160 mmHg, or diastolic blood pressure ≥100 mmHg), etc.).
18. Uncontrolled diabetes (defined as HbA1c>10.0%).
19. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) is more than twice the upper limit of normal (ULN), and/or serum creatinine is 1.2 times more than the ULN, and is clinically significant in the opinion of the Investigator.
20. Abnormal coagulation function（prothrombin time ≥ 3 seconds over ULN, activated partial thromboplastin time ≥ 10 seconds over ULN）
21. Active disseminated intravascular coagulation and obvious bleeding tendency within 3 months prior to dose 1.
22. Evidence of significant uncontrolled concomitant diseases such as cardiovascular diseases, nervous system diseases, respiratory system diseases, urinary system diseases, digestive system diseases and endocrine diseases.
23. Current treatment for active systemic infection, or history of recurrent serious infections.
24. Known active or suspected autoimmune diseases, requiring systemic immunosuppressive therapy.
25. Positive for syphilis screening test or positive for human immunodeficiency virus (HIV) screening test.
26. Known allergy to any component of the study intervention or history of allergy to fluorescein or indocyanine green, any anesthetics or antimicrobial agents used during the course of the study.
27. In the Investigator's judgment, other conditions considered not amenable to this study.
28. Participant who has been diagnosed to be COVID-19 or who has received COVID-19 vaccine within 1 month prior to dose 1.

Other protocol defined inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
Mean change of letters from baseline in best-corrected visual acuity (BCVA) at Week 48. | from baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

SECONDARY OUTCOMES:
Mean change of letters from baseline in the BCVA over time | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Proportion of patients gaining at least 15/10/5 letters in the BCVA at Week 12, 24, 36 and 48 | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Mean change from baseline in the total area of CNV and the total area of fluorescein leakage on fluorescein angiography (FA) at Week 12, 24 and 48 | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Mean change from baseline in central retina thickness (CRT) on optical coherence tomography (OCT) at Week 12, 24, 36 and 48 | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Change from baseline in National Eye Institute Visual Functioning Questionnaire - 25 scale score at Week 12, 24, and 48 | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Percentage and severity of ocular AEs (IVT procedure related and Investigation Medication related), non-ocular AEs; laboratory abnormalities; vital sign, physical examination abnormalities, etc. | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Incidence of ADAs and NAbs against HLX04-O following IVT administration | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
HLX04-O serum concentrations before Dose 1, Dose 2, Dose 6, Dose 9 and Dose 12 and the last visit as data permit. | From baseline to week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

CONTACTS AND LOCATIONS:
Locations (41):
- China (41):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Third Military Medical University (Southwest Hospital), Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Affiliated Hospital of Jinan University (Guangzhou Overseas Chinese Hospital ), Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanjing, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First People's Hospital of Zunyi, Zunyi, Guizhou
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Luoyang Third People's Hospital, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical College, Xinxiang, Henan
  - Henan Eye Hospital, Zhengzhou, Henan
  - People's Hospital of Wuhan University (Hubei Provincial People's Hospital), Wuhan, Hubei
  - Tongji hospital, Tongji medical college, Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan AIER Eye Hospital, Wuhan, Hubei
  - Wuhan Puren Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Affiliated Eye Hospital of Nanchang University, Nanchang, Jiangxi
  - the First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Hospital of Jilin University, Jilin, Jilin
  - Shenyang AIER Eye Hospital, Shenyang, Liaoning
  - Ningxia Hui Autonomous Region Peoples Hospital, Yinchuan, Ningxia
  - Shangdong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang Eye Hospital, Weifang, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - Zhejiang provincial people's hospital, Hangzhou, Zhejiang
  - Lishui Municioal Central Hospital, Lishui, Zhejiang

IPD SHARING:
Plan to Share IPD: No